CLINICAL TRIAL: NCT02075242
Title: Open Label, Multi-center, Randomized Study to Compare of Tacrolimus and Steroids in Combination With Mycophenolate Mofetil or Without Mycophenolate Mofetil in Liver Transplantation With Hepatitis B Virus(HBsAg) Positive
Brief Title: TO Compare the Triple Drug Therapy and Dual Therapy .
Acronym: OPTIMUS-A
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Gyu Lee, Professor, Department of surgery, Asan medical center, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0900; 2011-0900 (Other: ASAN MEDICAL CENTER Institutional review board)
Record Dates: First submitted 2014-02-26; First posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: HEPATITIS
Keywords: HBV
MeSH Terms: conditions — Hepatitis | interventions — Mycophenolic Acid; Tacrolimus; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tacrolimus (Active Comparator): Control group: Tacrolimus + Corticosteroid (dual oral therapy)
  Interventions: Drug: Tacrolimus
- Mycophenolate Mofetil (Experimental): Tacrolimus + Mycophenolate Mofetil+Corticosteroid (triple oral therapy)
  Interventions: Drug: Mycophenolate Mofetil; Drug: Tacrolimus

INTERVENTIONS:
Drug: Mycophenolate Mofetil — experimental group receive Tacrolimus as a main immunosuppressants and assistant is My-rept capsule®(Mycophenolate Mofetil),
  Other Names: Tacrolimus + Mycophenolate Mofetil+Corticosteroid
  Arms: Mycophenolate Mofetil
Drug: Tacrolimus — control group receive same immunosuppressants except for My-rept capsule®(Mycophenolate Mofetil- investigational product
  Other Names: Tacrolimus + Corticosteroid

SUMMARY:
Study to Compare the Safety and Efficacy of Tacrolimus and Steroids in Combination With Mycophenolate Mofetil or Without Mycophenolate Mofetil in Liver Transplantation with Hepatitis B Virus(HBsAg) Positive

ELIGIBILITY:
Inclusion Criteria:

* Men or women at the age of 20 to 65

  * Patients who will have primary Liver Transplantation becaused of Chronic Hepatitis B of HbsAg positive

    * Having confirmed a result of HBsAg positive patients within 6 months prior to Screening point.

      * Patients who will have Liver Transplantation from ABO-compatible or proper living donor ⑤ Patients who will receive investigational products for the entire period of clinical trial.

        * Patients who have signed the informed consent after understanding of clinical trial's purpose and risk.

          * For women of childbearing potential, pregnancy test negative from urine or blood AND women who agree to contraception for the entire period of clinical trial.

Exclusion Criteria:

* Recipients who had Liver Transplantation OR who had or will have other organ transplantation

  * Recipients who other organ transplantation in addition to liver at once.

    * Recipients who will have Auxiliary Partial Orthotopic Liver Transplantation.

      * Recipients who use a Bioartificial liver prior to Transplantation

        * Cr > 2.0mg/dl at screening test

          * Patients who had malignant tumor within the past 5 years OR have malignant tumor(except, successfully treated Skin's non-metastatic basal cell carcinoma, squamous cell carcinoma or primary hepatocellular carcinoma )

            * Recipients had hepatocellular carcinoma whick is out of Milan criteria

              * WBC<1,500/mm3 or ANC<900/mm3 or PLT<30,000/mm3 at Screening

                * Investigator judge that a patient is not proper to enroll this study due to Severe digestive disorder at Screening

                  * Patients who have severe systemic infection (But the liver transplantation is excepted that performed after the infection is completely lost or well-controlled)

                    ⑪ Recipients who had Liver transplantation from HBsAg positive donor

                    ⑫ Recipients or Donors are HIV, HCV Positive

                    ⑬ Patients who need to systemc chemotherapy or immunosuppressive therapy prior to transplantation or took immunosuppressants within 30 days prior to liver transplantation(except, investigational products per protocol and corticosteroid)

                    ⑭ Patients who have hypersensitivity to mycophenolate, mycophenolate acid, ingredient of investigational products, tacrolimus , Macrolide antibiotic and Steroids

                    ⑮ Patients who had been received or have been received other investigational products within 28 days prior to screening 16 Pregnant women and lactating women 17 Substance abuse patient, mentally defective person or patients who is not possible to participate in clinical trial by law 18 Investigator judge that a patient have communication disorder 19 Patients are not capable of visiting accor.ding to study visit schedule 20 Investigator judge that a patient is not proper to enroll this study, et cetera

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
rejection | within 6months
  • Incidence rate has been confirmed acute cellular rejection(RAI 4 and over) from liver biopsy

SECONDARY OUTCOMES:
rate of HBV | within 6 months
  • Recurrence rate of HBV after liver transplantation for 24 weeks (HBsAg Positve)
Graft survival rate | within 6 months
  • Patients survival rate after liver transplantation for 24 weeks / Graft survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Gyu Lee, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Korea, South Korea